CLINICAL TRIAL: NCT04657731
Title: Do Sociodemographic Factors Affect Occupational Balance?
Brief Title: Sociodemographic Factors and Occupational Balance
Acronym: SF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İnal, principal investigator, Hacettepe University
Other Study IDs: 06/11
Record Dates: First submitted 2020-12-02; First posted 2020-12-08 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-09

CONDITIONS: Occupational Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Occupational balance is a concept related to health and well-being. Therefore, determining the factors affecting this concept is important for health promotion interventions. There is no study in the literature on the relationship between socio-demographic factors and occupational balance. The results of this study are thought to provide new information to the literature.

DETAILED DESCRIPTION:
Occupational balance is about the perception of having the 'right mix' of activities in life. This balance is analyzed according to types of activity such as self-care, productivity and leisure time, as well as different dimensions such as the physical, mental and social dimensions required to engage in activities. Occupational balance is a concept related to health and well-being. Therefore, determining the factors affecting this concept is important for health promotion interventions. There is no study in the literature on the relationship between socio-demographic factors and occupational balance. The results of this study are thought to provide new information to the literature.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 19-70 Agree to participate in the study

-

Exclusion Criteria:

<19 years of age, >70 years of age

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals aged 19-70
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-12-09 (Estimated); Study Completion 2020-12-09 (Estimated)

PRIMARY OUTCOMES:
Occupational Balance Questionnaire Balance Questionnaire (OBQ11-T) | 3 months
  The OBQ is a scale that measures self-rated occupational balance in different dimensions.It contains 11 items and 4 response categories.Each item in the scale is scored on a 4-point scale from 'strongly disagree' to 'strongly agree'. The total score is obtained by summing the individual items and ranges from 0 to 33, with higher scores indicating higher occupational balance.

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)